CLINICAL TRIAL: NCT05621356
Title: Monitoring Allergen Immunotherapy in Allergic Rhinitis; is Nasal Fluid the Way to Precision Medicine?
Brief Title: Monitoring Allergen Immunotherapy in Allergic Rhinitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rijnstate Hospital (Other)
Collaborators: Wageningen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-1924; NL78278.091.21 (Other: CCMO)
Record Dates: First submitted 2022-11-10; First posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Immunotherapy; Rhinitis, Allergic; Treatment Outcome
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- allergen-specific immunotherapy (AIT): Adults with birch pollen allergy, who are treated with allergen-specific immunotherapy (AIT)
  Interventions: Other: A nasal fluid Basophil Activation Test (BAT)
- control: Adults with birch pollen allergy, who are treated with immunosuppressive medication
  Interventions: Other: A nasal fluid Basophil Activation Test (BAT)

INTERVENTIONS:
Other: A nasal fluid Basophil Activation Test (BAT) — a BAT technique for monitoring the inhibitory effect of nasal fluid on basophil activation.

SUMMARY:
Allergic rhinitis (hay fever) can be treated successfully with allergen-specific immunotherapy (AIT) for 3-5 years. This relative expensive and prolonged treatment is not suitable for everyone and therefore it is important to predict who will benefit from this therapy early after the start of treatment.

This project will investigate whether a BAT with nasal fluid can detect inhibition during immunotherapy in comparison with a BAT with blood.

DETAILED DESCRIPTION:
Allergic rhinitis (hay fever) can be treated successfully with allergen-specific immunotherapy (AIT) for 3-5 years. This relative expensive and prolonged treatment is not suitable for everyone and therefore it is important to predict who will benefit from this therapy early after the start of treatment. Biomarkers, like Basophil Activation Test (BAT) and IgE-facilitated allergen binding (FAB), using nasal fluid instead of blood, probably better reflect therapy effect (inhibition of an IgE-mediated allergic reaction) as the nose is the main target organ for AIT in allergic rhinitis.

This project will investigate whether a BAT with nasal fluid can detect inhibition during immunotherapy in comparison with a BAT with blood. Nasal fluid and blood samples are collected at baseline and after 8 and 16 weeks of treatment. A nasal fluid inhibition BAT is developed and validated by comparison with a BAT using serum and an IgE-FAB assay.

15 adults with birch pollen allergy, who are treated with AIT (Itulazax birch pollen tablet) and 10 adults with birch pollen allergy, who are treated with immunosuppressive medication (control group) will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* IgE-sensitized birch pollen allergy
* Start of Itulazax therapy or immunosuppressive therapy (nasal corticosteroid and/or antihistamine eye drops)
* Signed informed consent

Exclusion Criteria:

* Other underlying chronic conditions (immunological (autoimmune or immunodeficiency), oncological)
* Unstable uncontrolled asthma
* Smoking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Birch pollen allergic patients who are treated with Itulazax (birch pollen SLIT-tablet) and birch pollen allergic patients who are treated with immunosuppressive medication (control group).
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2022-12-23 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
BAT outcome nasal fluid | 8 weeks
BAT outcome nasal fluid | 16 weeks
BAT outcome serum | 8 weeks
BAT outcome serum | 16 weeks

SECONDARY OUTCOMES:
IgG4/IgA-associated inhibitory activity in nasal fluid | 8 weeks
IgG4/IgA-associated inhibitory activity in nasal fluid | 16 weeks
IgG4/IgA-associated inhibitory activity in serum | 8 weeks
IgG4/IgA-associated inhibitory activity in serum | 16 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Rijnstate Hospital, Arnhem, Netherlands